CLINICAL TRIAL: NCT00633698
Title: Evaluation of the Effect of NICOtinic Acid (Niacin) on Elevated Lipoprotein(a) Levels (NICOLa Study)
Acronym: NICOLa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. Elisabeth Steinhagen-Thiessen, Charité University Medical Center, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ep_Li 001_2006; EudraCT No.: 2006-005710-12
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Elevated Lipoprotein(a) Levels
Keywords: lipoprotein(a); niacin; placebo; intervention
MeSH Terms: interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Nicotinic acid (niacin)
  Interventions: Drug: Nicotinic acid (niacin)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinic acid (niacin) — oral medication Week 1-4: 500 mg per day Week 5-8: 1000 mg per day Week 9-12: 1500 mg per day Week 13-20: 2000 mg per day
  Other Names: Niaspan
  Arms: 1
Drug: Placebo — Placebo Week 1-4: 500 mg per day Week 5-8: 1000 mg per day Week 9-12: 1500 mg per day Week 13-20: 2000 mg per day
  Arms: 2

SUMMARY:
Lipoprotein (Lp)(a) has been associated with increased risk of cardiovascular disease. Niacin has been shown to lower Lp(a) in patients with normal or moderately elevated levels. However, there are few studies assessing the effectiveness of niacin in Lp(a) levels above 30 mg/dl. In addition, most studies investigating the effectiveness of niacin have only included small numbers of patients. Also, Lp(a) was only assessed as a secondary endpoint. The aim of the present study was, therefore, to evaluate whether Niacin is effective compared to placebo in the reduction of an elevated Lp(a).

DETAILED DESCRIPTION:
The study is a randomised, multicentre, placebo-controlled, 2-arm, parallel group, phase III, intervention study. Following randomisation at visit 1, subjects will receive 20 weeks of treatment with niacin or placebo.

The research question is: niacin therapy effective in lowering elevated Lipoprotein (Lp)(a) levels in comparison to placebo?

Sample size calculation is based on the t test of equal means with unequal group size (ratio: treatment group / control group = 2:1). The significance level is α=0.05 and the power 90%. Assuming a drop-out rate of 20%, sample size is 100 in the niacin group and 50 in the placebo group.

The active ingredient in the modified (prolonged, extended) release tablets is nicotinic acid, a B-complex vitamin. Modified release tablets containing 500 mg nicotinic acid, once daily for oral use, will be used.te of 20%, sample size is 100 in the niacin group and 50 in the placebo group.

Subjects will be recruited consecutively in the participating lipid clinics.

Subjects will be assessed at week -4 (run-in / wash-out), 0a+b (screening phase), 1, 5, 9, 13, and 20. Descriptive statistics will be used to summarize continuous and categorical variables. Mean change of Lp(a) levels will be compared between treatment and placebo group. Subjects will be grouped according to treatment randomised (intention-to-treat, ITT population). For missing data, the last observation will be carried forward (LOCF). Comparisons between groups will be performed using analysis of covariance (ANCOVA) with treatment as a factor, adjusting for baseline Lp(a) levels and other potential confounders.

Subgroup analyses will be performed according to Lp(a) phenotype, Lp(a) baseline level ( > 30-60 mg/dl, > 60 mg/dl), and concurrent statin therapy (yes / no).

Risks:

Flushing is the most common side effect of niacin. Other side effects include gastrointestinal disorders (common) (diarrhoea, nausea, vomiting, abdominal pain, or dyspepsia) and cardiac disorders (uncommon) (tachycardia, palpitations). A reversible elevation of liver enzymes has been reported, as well as a decreased glucose tolerance, reductions in platelet counts, increases in prothrombin time, elevations in uric acid levels, and reductions in phosphorous levels (uncommon or rarely). Hypersensitivity reactions have been reported very rarely.

Single reports on rhabdomyolysis in patients on combined therapy with niacin and HMG-CoA reductase inhibitors (statins) have been reported. Careful monitoring for any signs and symptoms of myopathy such as muscle pain, tenderness, or weakness is therefore required in the case of combination therapy.

Benefit:

Niacin has been shown to improve the lipid profile in patients with reductions in total cholesterol, LDL cholesterol and triglycerides and increases in HDL cholesterol. Niacin may also reduce elevated Lp(a) levels and may thus lower cardiovascular events in the long term.

The following variables will be assessed prior randomisation: socio-demographic factors, physical examinations, medical history, concurrent medication, health-related quality of life, costs prior study entry, and lipid as well as other laboratory parameters. Lipid parameters include Lp(a), total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides.

At follow-up, the respective laboratory analyses and physical examinations will be assessed at each visit. Subjects will be investigated with regard to safety and tolerability. Health-related quality of life and costs will be assessed at week 9 and 20.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 - 75 years
* Subjects with and without cardiovascular diseases
* Lp(a) plasma levels > 30 mg/dl
* Triglyceride levels < 400 mg/dl
* Cholesterol and triglyceride levels not requiring immediate change in medication according to current clinical guidelines
* If concurrent statin therapy, stable doses are required in the four weeks prior study inclusion, and no changes in statin dosages are allowed during the study period
* Subjects willing to follow all study procedures including attendance at practices for scheduled study visits, fasting prior to blood draws and compliance with study treatment regimen
* Written informed consent to participate in the trial

Exclusion Criteria:

* Known hypertriglyceridaemia or fasting triglycerides >= 400 mg/dl in the last four weeks before the randomisation visit.
* Known heterozygous or homozygous familial hypercholesterolaemia or known type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia)
* Documented secondary hypercholesterolaemia of any cause
* Initiation of a lipid-modifying drug treatment or a dose change of a lipid-modifying drug within the last four weeks
* Known hypersensitivity to nicotinic acid or any component of this medication or their derivatives
* Concurrent treatment with products containing significant amounts (more than 100 mg as daily dose) of nicotinic acid (niacin) or nicotinamide (e.g., vitamin preparations and nutritional supplements)
* Concurrent treatment with an immediate release formulation of nicotinic acid or a nicotinic acid analogue, e.g. supplements
* Treatment with an anticoagulant such as marcumar
* Cardiovascular diseases which are contra-indicated: unstable angina, acute myocardial infarction or uncontrolled cardiac arrhythmias within the preceding 3 months, stroke within the preceding 6 months, symptomatic heart failure (NYHA class III or IV), or severe peripheral artery disease
* Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception (prescription oral contraceptives, abstinence, condoms with spermicide, surgical sterilisation, diaphragm with spermicide, or intrauterine device)
* History of malignancy, except subjects who have been disease free for more than 10 years or whose only malignancy has been basal or squamous cell skin carcinoma. Women with a history of cervical dysplasia should be excluded unless 3 consecutive normal cervical smears have subsequently been recorded before entry into the study.
* History of alcohol (more than 2 glasses of wine or alcohol equivalent per day) or drug abuse (within 12 months of screening), or both
* Active liver disease or hepatic dysfunction as defined by elevations of AST or ALT >=1.5 times the ULN in the last 4 weeks before the randomisation visit
* Known uncontrolled or poorly controlled (HbA1C > 9 %) diabetes
* Persistent uncontrolled or untreated hypertension, defined as either resting diastolic blood pressure of > 95 mmHg or resting systolic blood pressure of > 200 mmHg
* Unexplained serum creatine phosphokinase (CK) > 3 times the ULN in the last 4 weeks before the randomisation visit (e.g. not due to recent trauma, intramuscular injections, heavy exercise etc)
* History of severe myalgia of unknown origin
* Arterial bleeding
* Active peptic ulcer
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Active gout symptoms
* Significant renal insufficiency (serum creatinine > 1.5 mg/dl)
* Planned hospitalizations for diagnostic or surgical procedures within the next 5 months
* Known infectious disease such as hepatitis or HIV
* Participation in another investigational drug trial within the four weeks prior to study entry
* Previous randomisation into this study
* Subjects with serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Persons who are detained officially or legally to an official institution.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Mean change in Lp(a) levels | 20 weeks

SECONDARY OUTCOMES:
Mean change in total cholesterol levels | 20 weeks
Mean change in LDL (low density lipoprotein) cholesterol levels | 20 weeks
Mean change in HDL (high density lipoprotein) cholesterol levels | 20 weeks
Mean change in triglyceride levels | 20 weeks
Mean change in blood glucose levels | 20 weeks
Health-related quality of life | 20 weeks
Disease-related costs | 20 weeks
Clinical adverse events | 20 weeks
Laboratory safety parameters | 20 weeks
Adherence to medication | 20 weeks
Tolerability of medication | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Steinhagen-Thiessen, MD, Study Director — Lipidambulanz und Lipidapherese, Charité Campus Virchow-Klinikum
Locations (1):
- Institute of Social Medicine, Epidemiology and Health Economics, Berlin, State of Berlin, Germany